CLINICAL TRIAL: NCT04327180
Title: PCR-COVID-19 Predictors of Positivity in Patients Admitted to ICU for Respiratory Infection: A Prospective Observational Cohort Study
Brief Title: PREdiction of DIagnosed Covid-19 infecTion in IUC Patients
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_20; 2020-A00763-36 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Infection Viral; Coronavirus; ARDS; Pneumonia
Keywords: critical care; biology of infectious agent
MeSH Terms: conditions — Virus Diseases; Coronavirus Infections; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients suspected of infection with COVID-19.: Patients included with positive PCR and patients with negative PCR included

SUMMARY:
Coronavirus 2019 (COVID-19) is a respiratory tropism virus transmitted through droplets emitted into the environment of infected persons. The symptoms can be extremely varied and the course can range from spontaneous healing without sequelae to death.

Currently, the diagnosis of certainty for resuscitation patients (by definition "severe") is based on searching for a fragment of virus genetic material within the epithelial cells of the respiratory tree, up and/or down, by PCR.

It is to be expected that the epidemic peak will make it difficult (if not impossible) to respect the stereotypical path that is currently in place, due to the lack of space in the specific unit. This will require optimization of care pathways and use of the specific sectors.

It is therefore necessary to define the simple criteria, available from the moment patients are admitted, to predict the result of the COVID-19 PCR.

ELIGIBILITY:
Inclusion Criteria:

* All patient admitted in ICU Lille Hospital and hospitalized in the unit "Emergent Biological Risk" (REB) before a suspicion of infection with COVID-19
* Clinical infectious syndrome: fever (>38°C) or hypothermia ( 36°C), chill, fever at home
* a severe respiratory table defined by:
* Oxygen demand > 3 L/min in the presence of significant comorbidity (pregnancy, chronic respiratory disease, chronic heart disease, hemopathy, cirrhosis) or > 6 L/min in the absence of comorbidity
* or a respiratory rate > 30 cycles per minute
* the need for mechanical, invasive or non-invasive ventilation
* the need for humidified high-flow oxygen therapy

Exclusion Criteria:

* Patient already included in study for first stay
* Cirrhosis CHILD C
* Major surgery in the last 7 days Minor patient
* Patient under guardianship or curatorship
* Refusal to participate
* No social security coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The selection of patients will be carried out by a Doctor of Medicine practising within the ICU Lille Hospital taking care of patients suspected of infection with COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Correlation between nasal and deep PCR positivity for Covid-19 patients performed and all predictors for Covid-19 patients performed within 24 hours of admission to ICU | within 24 hours of admission to ICU

SECONDARY OUTCOMES:
Coinfections | during ICU stay, up to 28 days
  Assessment of viral, bacterial, fungal and parasitic rate in confirmed and unconfirmed patients for COVID-19
Respiratory dysfunction requiring mechanical ventilation | during ICU stay, up to 28 days
  it will be reported the evolution of respiratory dysfunction in patients infected with COVID-19 admitted to ICU during their stay and requiring mechanical ventilation (during, Pao2/FIO2 ratio,,features of artificial ventilation features of extra-bodied respiratory assistance)
Sequential Organ Failure Assessment (SOFA) Score | during ICU stay, up to 28 days
  the SOFA assessment is used to track a person's risk status during stay in the Intensive Care Unit (ICU). The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal, and neurological systems. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure).
SAPS II score | at admission
  APS II was designed to measure the severity of disease for patients admitted to Intensive care units 24 hours after admission to the ICU, the measurement has been completed and resulted in an integer point score between 0 and 163 and a predicted mortality between 0% and 100%.
Disseminated Intravascular Coagulation (DIC) score | during ICU stay, up to 28 days
  The DIC Score was developed by the The International Society of Thrombosis and Haemostasis (ISTH.) The DIC score calculator accounts of the following four parameters.Each of the four parameters evaluated above have values that are weighted with a number of points varying from 0 to 3. By summing the points given to the choices, a final result between 0 and 8 is obtained
Number of days on vasopressive amines | during ICU stay, up to 28 days
Occurrence of an event of venous or arterial thromboembolic disease | during ICU stay, up to 28 days
Number of days with extra renal treatment (ERA) | during ICU stay, up to 28 days
Number of patients alive after ICU stay less than 28 days will be tracked | At 28 day
Short Form 36 | at 9 months +/- 3 months after ICU stay
  measuring the long-term impact of confirmed COVID-19 infection. assessment of quality of life according to 8 areas: physical activity (and related limitations), body pain, perception of one's own health, mental health (and related limitations), social life and vitality.
Hospital anxiety and depression scale (HADS) | at 9 months +/- 3 months after ICU stay
  The scale allows to detect anxiety and depression using 14 items rated from 0-3.
  Measuring the long-term impact of confirmed COVID-19 infection
Impact of Event Scale - revised (IES-R) | at 9 months +/- 3 months after ICU stay
  22-item self-report measure that assesses subjective distress caused by traumatic events Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88) Measuring the long-term impact of confirmed COVID-19 infection
Post-traumatic stress disorder Checklist version DSM-5 (PSL-5) | at 9 months +/- 3 months after ICU stay
  Question the stressful experience or event, followed by 20 multiple-choice questions.
  Measuring the long-term impact of confirmed COVID-19 infection
Modified Medical Research Council (MMRC) Dyspnea Scale | at 9 months +/- 3 months after ICU stay
  The mMRC Dyspnea Scale stratifies severity of dyspnea in respiratory diseases Measuring the long-term impact of confirmed COVID-19 infection
Correlation between number of patient deaths and all predictors for Covid-19 including anamnestic, clinical, biological, radiological parameters | until day 28 after admission of ICU
Viral clearance | through study completion, an average of 28 days
  Evolution of viral clearance in nasal and depp PCR during ICU

CONTACTS AND LOCATIONS:
Overall Officials: Julien Poissy, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, ICU, CHU Lille, Lille, France

REFERENCES:
- [Derived] Ledoult E, Guerrier T, Dubucquoi S, Figeac M, Villenet C, Daunou B, Behal H, Pokeerbux MR, Machet T, Koether V, Collet A, Launay D; Lille Covid Research network (LICORNE). Dual role of plasmablasts as immune regulators or amplifiers in COVID-19. Clin Immunol. 2025 Oct 13;281:110609. doi: 10.1016/j.clim.2025.110609. Online ahead of print. PMID 41093046